CLINICAL TRIAL: NCT03151330
Title: Serum Assessment of Preterm Birth: Outcomes Compared to Historical Controls
Brief Title: Serum Assessment of Preterm Birth Outcomes Compared to Historical Controls: AVERT PRETERM TRIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Principal Investigator, Matthew Hoffman, Chair Department of OB/GYN, Christiana Care Health Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DDD603819
Record Dates: First submitted 2017-04-22; First posted 2017-05-12 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Women who are found to have an elevated risk of preterm birth will receive counseling regarding potential interventions and compared to historical controls
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screened arm (Other): This will be an arm of women who are prospectively screened and receive a risk score for preterm birth. They will be recommended treatment strategies and their outcomes compared to an historical control.
  Interventions: Other: Screened Arm

INTERVENTIONS:
Other: Screened Arm — Woman who are identified as high risk will be advised of potential interventions which will include support through care link(nurse education), cervical surveillance, consider vaginal progesterone, low dose aspirin if not already taking.

SUMMARY:
Background: Preterm birth (PTB) remains the leading cause of neonatal mortality and long term disability throughout the world. Recently treatments early in pregnancy such as progesterone, cervical support and maternal support have been demonstrated to delay delivery amongst at risk women. Nonetheless, the majority of women who are at risk are not identified using current screening modalities.

Hypothesis: A cohort of pregnancies who are screened using the PreTRM® test around 20 weeks gestation in which a bundle of interventions is given for elevated PreTRM® risk will show either decreased neonatal morbidity/and mortality (measured as a composite score, "NMI"), or decreased length of neonatal stay in the hospital (NNOLOS). Secondarily, they will show an increase in gestational age at birth (GAB) and a reduction in length of neonatal NICU stay (NICULOS), compared to an unscreened historical control group.

Study Design Type: Prospective cohort study of screened women compared to a historical control of 10000 women.

DETAILED DESCRIPTION:
Population: Women who are 18 years or older, with a singleton pregnancy between 195/7 weeks and 206/7 weeks gestational age (GA) confirmed by ultrasound prior to enrollment, and no history of prior preterm birth (delivery between 160/7 weeks and 366/7 weeks) will be invited to participate. A comparable population will be identified using a historical control group in a contemporaneously maintained database.

Intervention: Qualifying women will be screened using the PreTRM® test (Sera Prognostics, Inc.) at a large tertiary care center. Predicated upon the degree of risk, women will be treated according to a prespecified algorithm. The outcomes of these women will be compared to a historical control group at the same tertiary care center.

Outcomes:

Primary outcome: Co-Primary outcomes: To determine whether a cohort of women who are screened with the PreTRM® test and then managed according to a prespecified protocol will have statistically significant reductions in either (a) composite neonatal morbidity and mortality (NMI score), or (b) length of neonatal hospital stay (NNOLOS), compared to a historical control group. The NMI is defined below

DEFINITIONS OF COMPOSITE PERINATAL MORTALITY/NEONATAL MORBIDITY OUTCOME SCORES:

1) 0 to 4 scale without NICU: This score was derived as an ordinal scale based upon severity. The score was defined by the following: 0 = no events;

1. = one event for (RDS, BPD, grade III or IV IVH, PVL, proven sepsis, or NEC) and no perinatal mortality,
2. = two events and no perinatal mortality;
3. = three or more events and no perinatal mortality; 4=perinatal mortality.

2) 0 to 4 scale with NICU: This score was defined as the following: 0 = no events,

1. = one event for (RDS, BPD, grade III or IV IVH, PVL, proven sepsis, or NEC) or <5 days in the NICU, and no perinatal mortality;
2. = two events or between 5 and 20 days in the NICU, and no perinatal mortality;
3. = three or more events or >20 days in the NICU, and no perinatal mortality;
4. = perinatal mortality.

3) 0 to 6 scale without NICU: This score was defined as the following: 0 = no events;

1. = one event for (RDS, BPD, grade III or IV IVH, proven sepsis, or NEC) and no perinatal mortality,
2. = two events and no perinatal mortality;
3. = three events and no perinatal mortality;
4. = four events and no perinatal mortality;
5. = five events and no perinatal mortality;
6. = perinatal mortality.

4) Any morbidity or mortality event: (yes/no)

* Adapted from Hassan SS, et al. Ultrasound Obstet Gynecol 2011; 38:18-31 Supplementary Information

Secondary outcomes: To determine whether women who are screened with the PreTRM® test and then managed according to a pre-specified treatment algorithm will have a statistically significant reduction in proportion of any type of preterm births (spontaneous and indicated), the total length of hospital stay for spontaneous preterm births, and total length of hospital stay for any preterm birth.

Observations:

* Neonatal death and stillbirth
* Birth weight and number of subjects with birth weight <1500g and <2500g
* Total number of days spent in the NICU and nursery
* Composite neonatal morbidity score and components
* Whether or not received surfactant
* Occurrence of pneumonia
* Number of days of mechanical ventilation
* Number of subjects with 5 minute Apgar < 7
* Occurrence of asphyxia
* Number of preterm deliveries at <37, <35 and <32 weeks
* Occurrence of preeclampsia
* Proportion of primiparous women experiencing preterm birth and spontaneous preterm birth
* NICU days for spontaneous preterm birth in primiparous women in prospective treatment arm are significantly less than NICU days in primiparous women in the control group of sPTB
* Correlation of blood levels of 17-OHPC and other progestin levels to outcomes and observations

General Outcomes:

Total cost of hospital care for both the mother and fetus beginning at initiation of care through primary delivery and 28 days of life.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older
* Singleton intrauterine pregnancy
* No medical contraindications to continuing pregnancy
* Subject has no signs and/or symptoms of preterm labor and has intact membranes
* Planned delivery at Christiana Care Health System,
* English speaking as consents from other languages will not be provided.

Exclusion Criteria:

* Women who have taken or plan to take progesterone beyond 14weeks gestation prior to study enrollment
* Previous history of sPTB less than37 weeks gestation or PPROM less than34 weeks gestation
* Multiple gestations-including a pregnancy that is now a single fetus due to a reduction procedure, vanishing twin, etc
* Known fetal genetic anomalies that are incompatible with life. Examples would include trisomy 13 and trisomy 18. Others would be left to the discretion of the site investigators
* Any other medical conditions that may be considered a contraindication per the judgment of the site investigator
* The subject has a planned cesarean section or induction of labor prior to 370/7 weeks of gestation
* The subject has a planned cerclage placement for the current pregnancy
* Major structural anomalies that may shorten pregnancy- examples would include anencephaly, holoprosencephaly, schizencephaly, gastroschisis, omphalocele, congenital diaphragmatic hernia, pyloric stenosis, etc. Minor anomalies such as polydactyly, unilateral hydronephrosis are not viewed as exclusions. Others would be left to the discretion of the site investigators
* History of cervical conization
* The subject has a uterine anomaly, History of classical cesarean section in a previous pregnancy
* The subject has had a blood transfusion during the current pregnancy
* The subject has known elevated bilirubin levels (hyperbilirubinemia)
* Previously identified short cervix (< 2.5 cm by TVUS)
* The subject has taken or plans to take any of the following medications after the first day of the last menstrual period: Enoxaparin, heparin, heparin sodium, low molecular weight heparin or the subject has a history of allergic reaction to aspirin or progesterone.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — requires pregnancy
Enrollment: 1873 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Neonatal Mortality Index | Birth through 6 months
  Outcomes:
  Co primary outcomes will consist of the Neonatal Morbidity Index as defined by Hassan and Neonatal NICU length of stay
Neonatal NICU length of stay | Birth to 6 months
  Duration of hospitalization in the NICU

SECONDARY OUTCOMES:
Preterm birth | Through pregnancy completion, typically 42 weeks
  Preterm birth before 37 weeks
Total length of hospital stay for any preterm birth | From birth to 60 days post delivery
  Total length of hospital stay for any preterm birth

OTHER OUTCOMES:
Neonatal death and stillbirth | Through 42 days post delivery
  Neonatal death and stillbirth
Birthweight and if birthweight was <1500g | At time of delivery
  birthweight below 1500 and 2500gm
Birthweight and if birthweight was <2500gm | At time of delivery
  birthweight below 2500gm
Whether or not received surfactant and amount of surfactant | Through hospitalization or 60 days post delivery
  Whether baby got surfactant
Occurrence of pneumonia | Through hospitalization or 60 days post delivery
  Occurrence of pneumonia
Number of days of mechanical ventilation | Through hospitalization or 60 days post delivery
  days on mechanical ventilation
Occurrence of 5 minute Apgar<7 | At time of birth
  low apgar as defined
Occurrence of asphyxia, diagnosed either via intrapartum cord gas or via clinical findings | At tiem of birth
  Occurrence of asphyxia,
Occurrence of preterm delivery at <37, <35 and <32 weeks | At time of birth
  Occurrence of preterm delivery at <37, <35 and <32 weeks
Occurrence of preeclampsia | Through 60 days post delivery
  preeclampsia as defined by ACOG
Progesterone levels determined by LC-MS | at 32 weeks
  progesterone levels

CONTACTS AND LOCATIONS:
Overall Officials: Matthew K Hoffman, MD, Principal Investigator — ChristianaCare
Locations (1):
- Christiana Hospital, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will potentially be shared with a like study being conducted at the University of Utah

REFERENCES:
- [Background] Anderson RN, Smith BL. Deaths: leading causes for 2001. Natl Vital Stat Rep. 2003 Nov 7;52(9):1-85. PMID 14626726
- [Background] Berghella V, Rafael TJ, Szychowski JM, Rust OA, Owen J. Cerclage for short cervix on ultrasonography in women with singleton gestations and previous preterm birth: a meta-analysis. Obstet Gynecol. 2011 Mar;117(3):663-671. doi: 10.1097/AOG.0b013e31820ca847. PMID 21446209
- [Background] CLASP: a randomised trial of low-dose aspirin for the prevention and treatment of pre-eclampsia among 9364 pregnant women. CLASP (Collaborative Low-dose Aspirin Study in Pregnancy) Collaborative Group. Lancet. 1994 Mar 12;343(8898):619-29. PMID 7906809
- [Background] Esplin MS, Elovitz MA, Iams JD, Parker CB, Wapner RJ, Grobman WA, Simhan HN, Wing DA, Haas DM, Silver RM, Hoffman MK, Peaceman AM, Caritis SN, Parry S, Wadhwa P, Foroud T, Mercer BM, Hunter SM, Saade GR, Reddy UM; nuMoM2b Network. Predictive Accuracy of Serial Transvaginal Cervical Lengths and Quantitative Vaginal Fetal Fibronectin Levels for Spontaneous Preterm Birth Among Nulliparous Women. JAMA. 2017 Mar 14;317(10):1047-1056. doi: 10.1001/jama.2017.1373. PMID 28291893
- [Background] Rittenberg C, Newman RB, Istwan NB, Rhea DJ, Stanziano GJ. Preterm birth prevention by 17 alpha-hydroxyprogesterone caproate vs. daily nursing surveillance. J Reprod Med. 2009 Feb;54(2):47-52. PMID 19301566
- [Background] Saade GR, Boggess KA, Sullivan SA, Markenson GR, Iams JD, Coonrod DV, Pereira LM, Esplin MS, Cousins LM, Lam GK, Hoffman MK, Severinsen RD, Pugmire T, Flick JS, Fox AC, Lueth AJ, Rust SR, Mazzola E, Hsu C, Dufford MT, Bradford CL, Ichetovkin IE, Fleischer TC, Polpitiya AD, Critchfield GC, Kearney PE, Boniface JJ, Hickok DE. Development and validation of a spontaneous preterm delivery predictor in asymptomatic women. Am J Obstet Gynecol. 2016 May;214(5):633.e1-633.e24. doi: 10.1016/j.ajog.2016.02.001. Epub 2016 Feb 11. PMID 26874297
- [Background] Romero R, Conde-Agudelo A, El-Refaie W, Rode L, Brizot ML, Cetingoz E, Serra V, Da Fonseca E, Abdelhafez MS, Tabor A, Perales A, Hassan SS, Nicolaides KH. Vaginal progesterone decreases preterm birth and neonatal morbidity and mortality in women with a twin gestation and a short cervix: an updated meta-analysis of individual patient data. Ultrasound Obstet Gynecol. 2017 Mar;49(3):303-314. doi: 10.1002/uog.17397. PMID 28067007

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT03151330/SAP_002.pdf